CLINICAL TRIAL: NCT03226860
Title: Improving Gait and Balance in Children With Hemiplegic Cerebral Palsy: Gait Myoelectric Stimulator Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.15
Record Dates: First submitted 2017-04-14; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait Myoelectric Stimulator (Experimental): The Gait Myoelectric Stimulator device stimulates the dorsiflexor and plantarflexor muscles at the correct time for typical walking.
  Interventions: Device: Gait Myoelectric Stimulator
- Ready, Set, Go! 5210 program (Active Comparator): Nationwide Initiative which recommends eating 5 servings a day of fruits and vegetables, 2 hours a day or less of screen time, 1 hour/day or more of physical activity, and 0 sugary drinks/day. This program supports the current focus in pediatric physical therapy on life-long fitness in youth with disabilities.
  Interventions: Other: 5210

INTERVENTIONS:
Device: Gait Myoelectric Stimulator — Electrical stimulation during gait for children with CP
  Other Names: GMES
  Arms: Gait Myoelectric Stimulator
Other: 5210 — Children will eat 5 fruits/vegetables each day, watch 2 hours or less of screen time, perform 1 hour or more of physical activity, and drink 0 sugar-sweetened beverages.
  Arms: Ready, Set, Go! 5210 program

SUMMARY:
This research study will see if electrical stimulation increases heel strike (heel hits the floor first when walking), decreases limp, helps muscle contraction, and improves balance in children with a hemiplegic leg. An experimental electrical stimulation device called the Gait MyoElectric Stimulator (GMES) will be used to stimulate the shin and calf muscles.

DETAILED DESCRIPTION:
Physical therapists focus on improving gait and balance in children with hemiplegic cerebral palsy (HCP). Functional electrical stimulation (FES) has the potential to improve strength and functional gait for children with HCP. The investigators hypothesize that a new FES system stimulating the dorsiflexor (DF) and plantarflexor (PF) muscles alternately at the correct time during gait, would lead to a significant improvement (p<.05) in foot contact, gait symmetry and balance, compared to 12 weeks of a healthy lifestyle program called 5210.

ELIGIBILITY:
Inclusion Criteria:

* Children who are:

  1. Are age 5-18 years
  2. Have been walking independently (no walker or cane) for at least 18 months.
  3. Use co-contraction of DF and PF during walking based upon surface electromyography.
  4. Have a diagnosis of spastic hemiplegic CP, Gross Motor Function Classification System (GMFCS) Levels I-II

Exclusion Criteria:

* Children who:

  1. Have passive ankle range <5 DF or < 10 PF with hip and knee extended.
  2. Report uncontrolled seizures.
  3. Had orthopedic surgery (for example heel cord or hamstring lengthening)
  4. Have used tone reducing medications (Botox, Baclofen) in the last 6 months.
  5. Wear ankle foot orthoses that limit DF/PF motion.
  6. Have low motivation/tolerance for electrical stimulation.
  7. Have parents/caregivers who are not able or willing to assist with the protocol for 6 months.
  8. Have low tolerance to electrical stimulation in screening process.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Aim 1 - Improve initial contact during gait, as measured by Noraxon video software | 12 weeks
  To determine if the GMES program will improve initial contact during free speed walking (ie decrease toe first or flat foot contact, and increase heel strike).
  Based on visual examination of freeze frame videotaped walking patterns, "foot contact" will be scored at initial contact as either heel, foot flat, or toe. A numerical assignment will be placed for each of these contact points. Each step with the heel contact (the most optimal), will receive a score of 3. Each step with the foot flat (the less optimal), will receive a score of 2. Each step the toe contact, (the least optimal), will receive a score of 1. A total of 10 initial contacts will be examined at each testing. The numerical value of the total number of contact points will be calculated for each subject and each trial.

SECONDARY OUTCOMES:
Aim 2 - Improve walking symmetry, as measured by Noraxon video software | 12 weeks
  To determine if the GMES program will improve walking symmetry. Symmetry will be calculated using Noraxon for 10 strides for each testing. Normal walking consists of 60% of the time standing on one foot (stance phase) and 40% with the foot in the air (swing phase). It is common for children with hemiplegia to have asymmetrical stance between right and left legs.
  The stance phase begins when the foot makes contact with the ground (initial contact) and ends when the foot leaves the ground (toe-off). The swing phase begins with toe-off and ends at initial contact. These gait events (initial contact and toe-off) are determined from freeze frame videotape for children as they walk in the laboratory. Noraxon software calculates these times and determines the percentage for right and left leg.
  Gait symmetry will be assessed as the difference in the percentages of the stance phase for each subject.
Aim 3 - Improve balance, as measured by the Balance Subtest of the Bruininks-Oseretsky Test of Motor Proficiency (BOT2). | 12 weeks
  To Determine if the GMES program will improve balance skills based on the Balance Subtest of the Bruininks-Oseretsky Test of Motor Proficiency (BOT2). Balance will be measured on the unaffected and on the hemiplegic side using the Balance Subtest of the BOT2. This test assesses 9 balance areas:
  * Standing with feet apart on a line - eyes open,
  * Walking forward on a line,
  * Standing on one leg on a line - eyes open,
  * Standing with feet apart on a line - eyes closed,
  * Walking forward heel-to-toe on a line,
  * Standing on one leg on a line - eyes closed,
  * Standing on one leg on a balance beam - eyes open,
  * Standing heel-to-toe on a balance beam,
  * Standing on one leg on a balance beam - eyes closed. These balance activities are designed to become more difficult as they progress. They are scored based on how many seconds the subject can balance, or how many steps the subject takes on the balance beam. The total raw score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Brandsma, PT, DPT, PCS, Principal Investigator — Physical Therapist for Mary Bridge Children's Therapy at Good Samaritan

IPD SHARING:
Plan to Share IPD: Undecided